CLINICAL TRIAL: NCT06496932
Title: Management of Anxiety and Vital Signs With Music in Cesarean Delivery: A Randomized Controlled Trial
Brief Title: Music for Anxiety Management in Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Tuğba Dündar, Research Assistant, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Interventional trial
Record Dates: First submitted 2024-07-04; First posted 2024-07-11 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Pregnancy
Keywords: cesarean section; music; randomize trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Listen to music group (Experimental): The study group will be played music during the cesarean section.
  Interventions: Other: Listen to music
- Standart cesarean procedure (No Intervention): The control group continued to receive the routine care

INTERVENTIONS:
Other: Listen to music — Women in the intervention groups will listen to nature and bird sounds through over-the-ear headphones after spinal anesthesia for cesarean section until the suturing is completed.
  Arms: Listen to music group

SUMMARY:
A randomized controlled trial will be conducted to determine examine the effects of music played during cesarean delivery on maternal anxiety and vital signs.

DETAILED DESCRIPTION:
It will tested the hypotheses that there is no difference between the intervention and control groups of pregnant women after the intervention in terms of anxiety and vita lsymptoms.

ELIGIBILITY:
Inclusion Criteria:

- Aged between 18-35 years,

* Undergoing cesarean section under spinal anesthesia,
* Experiencing spontaneous and singleton pregnancy,
* With a gestational age greater than 37 weeks,
* Pregnant individuals who have had at least 4 routine check-ups during pregnancy conducted by a member of the research team,
* Scheduled for cesarean section (regardless of the number of previous cesarean sections).

Exclusion Criteria:

* Having high-risk pregnancies such as preeclampsia, early membrane rupture, and placental abruption, • Being scheduled for emergency cesarean section for any reason

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 32 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
anxiete level | 37th gestational weeks]
  State-Trait Anxiety Inventory: It can be applied to individuals over the age of 14. It consists of 20 items that determine how an individual feels at a certain moment and under certain conditions. The highest score that can be obtained from the scale is 80 and the lowest score is 20. The higher the calculated total anxiety score, the higher the anxiety level of the person filling out the inventory.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba Dündar, Study Chair — AydınAdnan Menderes University, Faculy of Nursing, Division Public Health Nursing
Locations (1):
- Adnan Menderes University, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request
Supporting Information: CSR
Time Frame: 6 months after publication
Access Criteria: relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.